CLINICAL TRIAL: NCT00500747
Title: A Phase I Randomized, Observer-Blinded, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Immunogenicity of Chiron Corporation's HCV E1E2/MF59 Vaccine Administered to Healthy HCV-Negative Adults
Brief Title: Chiron Corp HCV E1/E2 Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Director ORA, HHS/NIAID/DMID
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 01-002; 11806
Record Dates: First submitted 2007-07-12; First posted 2007-07-13 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Hepatitis C
Keywords: hepatitis C, HCV, vaccine, recombinant vaccine, adjuvant
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Group C: 100 mcg HCV E1E2/MF59 vaccine (Experimental): Sixteen subjects receive four doses of 100 mcg HCV E1E2/MF59 vaccine (0.5 mL total volume) and 4 subjects receive placebo at 0, 4, 24, and 48 weeks.
  Interventions: Biological: HCV E1E2/MF59; Drug: Placebo
- Group B: 20 mcg HCV E1E2/MF59 vaccine (Experimental): Sixteen subjects receive four doses of 20 mcg HCV E1E2/MF59 vaccine (0.5 mL total volume) and 4 subjects receive placebo at 0, 4, 24, and 48 weeks.
  Interventions: Biological: HCV E1E2/MF59; Drug: Placebo
- Group A: 4 mcg HCV E1E2/MF59 vaccine (Experimental): Sixteen subjects receive four doses of 4 mcg HCV E1E2/MF59 vaccine (0.5 mL total volume) and 4 subjects receive placebo at 0, 4, 24, and 48 weeks.
  Interventions: Biological: HCV E1E2/MF59; Drug: Placebo

INTERVENTIONS:
Biological: HCV E1E2/MF59 — The investigational vaccine contains envelope glycoproteins gpE1 and gpE2 and the adjuvant, MF59. MF59 is a sterile oil-in-water emulsion in a citrate buffer, which comprises 50 percent of the vaccine. The antigen and adjuvant are combined prior to the injection. The volume to be administered is 0.5 mL for all vaccine dose levels. The vaccine has a milky white opacity. Vaccine dosages: 4 mcg, 20 mcg and 100 mcg.
Drug: Placebo — Four doses sterile saline (0.5 mL total volume) at 0, 4, 24, and 28 weeks.

SUMMARY:
The purposes of this study are to evaluate the safety, tolerability, and effectiveness of a vaccine (the HCV E1/E2/MF59 vaccine) against hepatitis C (HCV). The vaccine will be given to 60 healthy adult volunteers (aged 18-45 years) and the study will compare the immune system (the body's protective response) response to the HCV E1/E2 vaccine given at different dosage levels: 4 micrograms, 20 micrograms, or 100 micrograms in MF59 adjuvant (substance that can improve vaccine effectiveness). The volunteers will be assigned randomly (by chance) to 1 of 4 different groups. Volunteers in each group will receive a shot of the vaccine or a placebo (shot with no medication). Participants will be involved in study related procedures for up to 71 weeks, which includes blood samples, recording symptoms on a diary card, and 4 vaccine or placebo injections.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) has emerged as a significant public health concern throughout the world. Its estimated prevalence in the US is 1.5 percent, or 2.7 million people with chronic infection. As many as 170 million people may have chronic HCV infection worldwide. The Centers for Disease control currently estimates that 40,000 HCV infections occur yearly in the US, with most current infection acquired through illegal injection drug use. It is estimated that 70 percent of those infected will develop chronic liver disease. The purpose of this study is to conduct a Phase I vaccine trial with a novel vaccine, HCV E1E2/MF59. The study objectives are to evaluate the safety, tolerability, and immunogenicity of HCV E1E2/MF59 vaccine administered to healthy adult subjects and to compare the immune response to HCV E1E2 vaccine given at 4, 20, or 100 mcg in MF59 adjuvant. Sixty healthy adults, aged 18-45, will be randomized to receive one of 3 different doses of vaccine or placebo. Each subject will receive vaccine at 0, 4, 24, and 48 weeks. Study procedures will include blood sample collections and questions regarding risk factors for acquiring HCV.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, hepatitis C virus (HCV) negative.
* 18-45 year old healthy adults. Insufficient data are available in adults to judge risk in children.
* In good general health as determined by medical history, physical examination and the following screening labs:
* Complete Blood Count (CBC): Total WBC (White Blood Cell): 3.5-14 thousand/microliter (MCL); Hemoglobin (Hgb): Men: 12.2-18 g/dl and Women: 10.5-17 g/dl.
* Creatinine: Men: less than or equal to 1.4 mg/dl; Women: less than or equal to 1.2 mg/dl.
* Glucose: 50 mg/dl to less than or equal to 109 mg/dl.
* Alanine Aminotransferase (ALT): Men 2-60 units/litre (U/I): Women: 3-40 U/I.
* Aspartate Aminotransferase (AST): Men: 2-50 U/I, Women 2-35 U/I.
* Total bilirubin: Men: less than or equal to 1.5 mg/dl: Women: less than or equal to 1.3 mg/dl.
* Urinalysis: negative or trace protein, negative glucose, less than or equal to 3 Red Blood Cells (RBC)/High Power Field (HPF) and less than or equal to 5WBC/HPF (in nonmenstruating females).
* Negative serum cryoglobulin
* Hepatitis B: negative Hepatitis B Surface Antigen (HBsAg) (using standard Food and Drug Administration FDA approved tests, e.g. Abbott or Organon).
* Hepatitis C: Anti-Hepatitis C Virus (HCV) negative and HCV Ribonucleic Acid (RNA) negative (using standard FDA approved tests, e.g. Abbott or Organon).
* HIV ELISA negative (using standard FDA approved tests, e.g. Abbott or Organon) (Written informed consent for HIV antibody testing will be obtained before obtaining the HIV sample.) Note: HIV vaccine volunteers who test positive by HIV ELISA and HIV western blot testing due to receipt of HIV vaccine may participate if they test negative by HIV DNA Polymerase Chain Reaction (PCR).
* Negative urine pregnancy test (females of child bearing potential) obtained at screening and at the day of each immunization.
* The ability to understand and sign a written informed consent document. Available for 16 months after the first injection so that follow-up may be completed.

Exclusion Criteria:

* Diabetes.
* Cancer other than squamous cell skin cancer which has been excised.
* History of myocardial infarction or arrhythmia requiring hospitalization.
* Syncope requiring hospitalization.
* Unconsciousness other than a simple concussion.
* Seizures other than febrile seizures as a child <5 years of age.
* Current liver disease (not including Gilbert's disease).
* Autoimmune disease (does not include thyroid disease or vitiligo).
* Splenectomy.
* Uncontrolled hypertension [blood pressure (BP) >150/90; anti-hypertensive medications are acceptable).
* Subjects with identifiable high-risk behavior for HCV infection as characterized by the following: injection drug use (IVDU) or cocaine snorting within the last year.
* Subject had a tattoo or body piercing within the past 6 months and/or is planning to acquire any tattoos or body piercing during the period of the study.
* Subjects with tattoos at the bilateral sites of needle insertion.
* Pregnant or lactating women. Women of child bearing potential must be using effective contraception for at least 30 days prior to initial immunization, unless for religious, social, or medical reasons they do not intend to have children and are practicing sexual abstinence. Subjects using birth control must agree to do so for the entire 64 week study period. Acceptable method of birth control is defined as hormonal contraceptives, intrauterine device (IUD), diaphragm with spermicide, condoms, a vasectomized partner or abstinence.
* Concomitant drug exclusion: corticosteroids (other than intranasal sprays or topical creams) or other known immunosuppressive drugs (such as chemotherapy for cancer); any experimental agent; any anti-tuberculosis medication, e.g., isoniazid (INH).
* Personnel engaged in the blinding of this study.
* Subjects who for any reason cannot adhere to the schedule of this protocol should not be enrolled in the study.
* Subjects who in the judgment of the investigator would not be good candidates due to medical, psychiatric, or social conditions which may interfere with or serve as a contradiction to adherence to the study protocol.
* Subjects with sex partners with known active Hepatitis B virus (HBV), HCV, or HIV infection.
* Currently abuses alcohol. Alcohol abuse is defined as requiring hospital admission for detoxification and therapy or alcohol use that has had a significant impact on personal relationships or ability to work productively.
* Not accessible by telephone or pager.
* Live attenuated immunization within 4 weeks of each vaccination.
* Inactivated immunization within 2 weeks of each vaccination.
* Febrile illness within 3 days of study entry based on verbal report by the subject.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2003-08; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety, tolerability, and immunogenicity of HCV E1E2/MF59 vaccine when administered at 3 dose levels on a multi-dose schedule. | Duration of study.

SECONDARY OUTCOMES:
Compare the immune response to HCV E1E2 vaccine given at 4 mcg, 20 mcg, or 100 mcg in MF59 adjuvant. | Weeks 0, 2, 4, 6, 8, 24, 26, 50, 52 and 64.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

REFERENCES:
- [Derived] Nguyen YTK, Chen F, Giang E, Saha S, Ueno LA, Chen C, Watson CT, Tzarum N, Wilson IA, Law M, Stanfield R. Structural and genetic signatures of two classes of HCV E2 neutralizing face antibodies from non-human primates immunized with a recombinant E1E2. bioRxiv [Preprint]. 2025 Oct 7:2025.10.07.680784. doi: 10.1101/2025.10.07.680784. PMID 41278834
- [Derived] Chen F, Nagy K, Chavez D, Willis S, McBride R, Giang E, Honda A, Bukh J, Ordoukhanian P, Zhu J, Frey S, Lanford R, Law M. Antibody Responses to Immunization With HCV Envelope Glycoproteins as a Baseline for B-Cell-Based Vaccine Development. Gastroenterology. 2020 Mar;158(4):1058-1071.e6. doi: 10.1053/j.gastro.2019.11.282. Epub 2019 Dec 4. PMID 31809725
- [Derived] Kachko A, Frey SE, Sirota L, Ray R, Wells F, Zubkova I, Zhang P, Major ME. Antibodies to an interfering epitope in hepatitis C virus E2 can mask vaccine-induced neutralizing activity. Hepatology. 2015 Dec;62(6):1670-82. doi: 10.1002/hep.28108. Epub 2015 Oct 16. PMID 26251214
- [Derived] Frey SE, Houghton M, Coates S, Abrignani S, Chien D, Rosa D, Pileri P, Ray R, Di Bisceglie AM, Rinella P, Hill H, Wolff MC, Schultze V, Han JH, Scharschmidt B, Belshe RB. Safety and immunogenicity of HCV E1E2 vaccine adjuvanted with MF59 administered to healthy adults. Vaccine. 2010 Aug 31;28(38):6367-73. doi: 10.1016/j.vaccine.2010.06.084. Epub 2010 Jul 7. PMID 20619382